CLINICAL TRIAL: NCT03769701
Title: Efficacy of Two Schemes of Self-monitoring Capillary Glucose to Monitor Glycemic Control in Mexican Women With GDM
Brief Title: Efficacy of Two Schemes of Self-monitoring Capillary Glucose in Gestational Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Perinatologia Isidro Espinosa de los Reyes (Other Government)
Responsible Party: Principal Investigator, ENRIQUE REYES-Munoz MD, Medical Science Researcher, Instituto Nacional de Perinatologia Isidro Espinosa de los Reyes
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017-1-53
Record Dates: First submitted 2018-12-06; First posted 2018-12-07 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1, SMGC four times/day (Active Comparator): Women with GDM and SMGC 4 times/day; fasting and 1-hour post-prandial of breakfast, lunch and dinner
  Interventions: Procedure: self-monitoring capillary glucose (SMCG)
- SMGC two times/day (Experimental): Women with GDM and SMGC 2 times/day; pre-prandial and 1-hour post-prandial of breakfast, lunch or dinner alternating the meal each day.
  Interventions: Procedure: self-monitoring capillary glucose (SMCG)

INTERVENTIONS:
Procedure: self-monitoring capillary glucose (SMCG) — To measure the capillary glucose with a glucometer according to the assigned group.

SUMMARY:
Gestational diabetes mellitus (GDM) affects 10 % of women who receive prenatal care at Instituto Nacional de Perinatología (Mexico, City). Currently, there is clear evidence on the utility of self- monitoring of capillary glucose (SMGC) to evaluate the efficacy of medical-nutrition therapy on glycemic control. However, the reports regarding the best pattern of SMGC in terms of frequency and number of determinations per day are limited. The objective of this study is to evaluate the efficacy of two SMGC schemes for monitoring glycemic control in Mexican women with GDM.

DETAILED DESCRIPTION:
Currently, the evidence from randomized clinical trials about the most appropriate scheme of SMGC for monitoring the glycemic control among women with GDM is limited. This study was designed to evaluate the efficacy of two different schemes of SMGC in GDM Mexican population, it is an open-label randomized clinical trial including 2 groups: group 1 (SMGC 4 times/day) measured in fasting and 1 hour postprandial of breakfast, lunch and dinner; group 2 (SMGC 2 times/day), measured preprandial and 1 hour postprandial, of breakfast, lunch or dinner, alternating the meal each day, from GDM diagnosis until the resolution of pregnancy. Additionally, determinations of insulin, lipids and glycosylated hemoglobin (HbA1c) will be determinate at enrollment, and between the 30-32 and 36-38 of gestation week. The primary outcome: To compare the proportion of women who achieve glycemic control using SMGC 4 times/day versus SMGC 2 times/day.

Secondary outcome: To compare the risk of new-born large for gestational age, gestational hypertension, preeclampsia, preterm birth, cesarean section, new-born weight, neonatal hypoglycemia, neonatal hyperbilirubinemia and entry to neonatal intensive care between groups. An analysis for intention of treatment will be made according to the recommendations of the CONSORT guidelines.

ELIGIBILITY:
Inclusion Criteria:

* GDM diagnosis, defined by 2 or more altered values during oral glucose tolerance test (75g-2h): Fasting ≥ 95 mg/dl, 1 hour ≥ 180 mg/dl and 2 hours ≥ 155 mg/dl.
* Singleton pregnancy between 12-32 weeks of gestation at GDM diagnosis.

Exclusion Criteria:

1. Multiple pregnancy.
2. Pregestational diabetes.
3. Fasting glucose > 126 mg/dl or random glucose > 200 mg/dl before 12 weeks of gestation.
4. Active pathology: systemic lupus erythematosus, rheumatoid arthritis, congenital or acquired cardiopathy, uterine leiomyoma > 10cm, renal insufficiency and chronic hypertension.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2018-12-07 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of women who achieve glycemic control. | from GDM diagnosis to delivery.
  Proportion of women with more than 80% of capillary glucose determination into the following goals: preprandial; 70 to 95 mg/dl and 1 hour post-prandial ≤ 140 mg/dl.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Perinatology, México, Mexico

IPD SHARING:
Plan to Share IPD: No